CLINICAL TRIAL: NCT07351747
Title: Effect of Laser Acupoints on Fallopian Tube Obstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hadeer Elsaid Abd-Elsalam Shalaby, Senior Physical Therapist, Kafrelsheikh General Hospital, Kafrelsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-711
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Laser; Acupoints; Fallopian Tube Obstruction
MeSH Terms: conditions — Fallopian Tube Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Group A) (Experimental): Patients will receive laser acupoints therapy addition to standard care.
  Interventions: Other: Laser acupoints therapy + Standard care
- Control Group (Group B) (Placebo Comparator): Patients will receive placebo laser acupoints therapy in addition to standard care.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Laser acupoints therapy + Standard care — Patients will receive laser acupoints therapy addition to standard care.
  Arms: Study Group (Group A)
Other: Standard care — Patients will receive placebo laser acupoints therapy in addition to standard care.
  Arms: Control Group (Group B)

SUMMARY:
This study aims to determine the efficacy of laser acupoint therapy on treating fallopian tube obstruction.

DETAILED DESCRIPTION:
Fallopian tube obstruction is a significant health concern that affects a substantial number of women worldwide, often leading to infertility and other reproductive issues. The fallopian tubes, essential components of the female reproductive system, play a crucial role in the process of conception by facilitating the transport of ova from the ovaries to the uterus.

The laser's focused light energy, when directed at specific acupoints linked to reproductive health, is hypothesized to activate the body's energy pathways or meridians, thereby facilitating healing and restoration of normal tubal function.

Although acupoint therapy shows promise, laser acupoint therapy offers potential advantages over traditional acupuncture by utilizing low-level lasers, which may enhance the treatment's efficacy. Laser acupoint therapy is noninvasive and painless, making it articularly appealing for patients who have a fear of needles or are sensitive to pain.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-35 years - nulliparous.
* Women diagnosed with fallopian tube obstruction.
* Body mass index less than 30 kg/m2.
* Consent to participate in the study.
* General good health with no major co-existing medical conditions that could interfere with the treatment or outcomes.
* No prior fertility treatments [e.g., In vitro fertilization (IVF), intrauterine insemination (IUI)] within the last 6 months.
* Ability to attend all scheduled sessions and follow-up assessments.

Exclusion Criteria:

* Currently pregnant or breastfeeding.
* History of pelvic surgery within the past year.
* Presence of severe systemic diseases such as active cancer or severe cardiovascular diseases.
* History of allergic reactions or adverse responses to acupuncture or laser therapies.
* Currently undergoing hormonal therapy or use of hormonal contraceptives.
* Current or recent history of genital tract infections, including sexually transmitted. infections, which could affect the reproductive system.
* Presence of significant uterine anomalies diagnosed through imaging that could impact fertility.
* Polycystic Ovary Syndrome (PCOS).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women diagnosed with fallopian tube obstruction.
Enrollment: 36 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Tubal patency | 3 months post-treatment
  Hysterosalpingography (HSG) will be used to assess tubal patency. It is a radiographic technique where a contrast material is injected into the uterine cavity, and X-ray images are taken to evaluate the shape of the uterus and the status of the fallopian tubes. HSG will be applied before the treatment and again three months post-treatment to evaluate changes in tubal patency HSG will be applied before treatment and after 3 months post-treatment.

SECONDARY OUTCOMES:
Anti-Müllerian Hormone (AMH) Test | 3 months post-treatment
  A blood test will be used to measure the level of Anti-Müllerian Hormone (AMH), which is an indicator of the remaining quantity of eggs and ovarian function. This test will be conducted before the treatment and at the third month of treatment to monitor any changes in ovarian reserve.
Quantitative Pregnancy Test | 3 months post-treatment
  A blood test that will be measured the specific level of Human Chorionic Gonadotropin (hCG), which is produced during pregnancy. This test will be performed every month.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University (Faculty of Physical Therapy), Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.